CLINICAL TRIAL: NCT01561625
Title: Signaling Pathway Activation in the Quadriceps of Patients With COPD After an Acute Bout of Resistance
Brief Title: Signaling Pathway Activation After Exercise in Patients With Chronic Obstructive Pulmonary Disease
Acronym: SIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Bruno Lemire, Étudiant au doctorat, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SIM-COPD-20458
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: exercise — resistance training exercise, 1 session, 3 exercises, 80% of max

SUMMARY:
Muscle weakness and atrophy are important consequences of chronic obstructive pulmonary disease (COPD). Although resistance exercises increase strength and muscle mass in patients with COPD, the response to training appears to be suboptimal in these individuals. A dysregulation in the signaling pathways involved in the regulation of muscle mass could play an important role in this phenomenon.

Hypothesis: Proteins involved in muscle mass regulation will be less activated in the quadriceps of patients with COPD following the acute bout of resistance training exercise compared to healthy age-matched controls.

DETAILED DESCRIPTION:
Our objective is to investigate the impact of an acute bout of resistance training on key signaling pathways involved in the regulation of muscle mass in moderate to severe COPD (FEV1 under 60% of predicted). Key proteins of signaling intramuscular pathways involved in protein synthesis and degradation will be measured before after 72 contractions of the quadriceps. The exercise protocol was designed to match the actual exercise prescription model use in the context of pulmonary rehabilitation. A squat, leg press and leg extension will be done at 80% of max with one minute rest between sets. A biopsy of the quadriceps will be done before and after exercise in order to measure phosphorylated kinases, total protein content and mRNA expressions. All our patients will undergo a thorough baseline assessment in pulmonary capacity, muscle force and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Male
* COPD with an FEV1 of under 60% of predicted
* non-smoker
* Between 50 and 75 years old

Exclusion Criteria:

* All inflammatory disease (HIV, Cancer, renal and cardiac deficiency)
* Hormonal dysregulation
* Inferior limb pathology
* Neuromuscular pathology
* History of tabacco or alcool abuse
* Oxygen dependent
* Recent exacerbation (2 months) of the symptoms of COPD

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Post-exercise signaling proteins phosphorylation level in the quadriceps of COPD patients and age-matched healthy controls | 2 hours post-exercise
  Phosphorylation status of key proteins (Akt, p70, mTOR, p38, JNK, ERK) will be lesser modulated in the quadriceps of patients with COPD compare to healthy controls. The phosphorylated as well as the total protein levels will be measured by western blot. The data will be presented as arbitrary units and compared with values obtained in healthy age-matched healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Laval University
Locations (1):
- IUCPQ, Québec, Quebec, Canada